CLINICAL TRIAL: NCT00155142
Title: Changes in Skin Innervation of Neurologically Asymptomatic Type 2 Diabetic Patients: the Correlation With the Diabetic Parameters and Neurotrophins.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701104
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2004-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To address the following issues: (1) the course of small nerve fiber degeneration in type 2 diabetic patients, especially in asymptomatic patients; (2) the influence of blood sugar control on development of the small fiber degeneration; (3) the correlation of skin innervation with sensory thresholds, autonomic tests and parameters of nerve conduction studies; and (4) the role of neurotrophins in diabetic neuropathy, we will perform skin biopsy with quantification of IENF in type 2 diabetic patient without neurological symptoms. The investigations all include clinical evaluation, electrophysiological studies, quantitative sensory test and enzyme linked immunosorbent assay of neurotrophins. The analysis of skin innervation with diabetic parameters will give important insights into the mechanism, prevention and management of small fiber neuropathy in neurologically asymptomatic type 2 diabetic patients, and also therapeutic strategies for diabetic neuropathy.

DETAILED DESCRIPTION:
Type 2 diabetes is one of the most common disorders in general population. The overall prevalence of type 2 diabetes among people older than 40 years old in Taiwan is about 10 %. Various complications are associated with diabetes and these complications have become an important issue in daily clinical practice.

Neuropathy is one of the most frequent symptomatic complications of diabetes and is potentially devastating. Small-fiber neuropathy is a major component of diabetic neuropathies and usually causes disabling symptoms like pain and burning. It typically begins at the distal limbs and progresses to the proximal part with time. Recent studies have indicated that skin innervation is reduced in neurologically symptomatic type 2 diabetic patients and the reduction is correlated with the duration of diabetes1. It is not clear whether similar changes occur in neurologically asymptomatic type 2 diabetes. Neurovascular disturbance (i.e. decreased skin blood flow) was noted in early and clinically silent diabetic patients and it might represent the functional and organic abnormalities in small unmyelinated C fibers. Along the same line it is reasonable to speculate that there might be changes in the skin innervation in the preclinical phase of diabetic neuropathic patients. No previous studies have investigated the course of the changes in skin innervation from early or asymptomatic stage to symptomatic stage in diabetic patients.

The relationship of diabetes and the occurrence of peripheral neuropathy had been studied by the Diabetes Control and Complications Trial Research Group and the Kumamoto study in type 1 or 2 diabetes respectively. The results showed that intensive control of hyperglycemia could prevent or delay the development of diabetic neuropathy. However the neuropathies in the studies were assessed by nerve conduction studies. These examinations are insensitive to the small fiber degeneration and it is not clear whether small fibers changes during intensive diabetic control. There is also lack of direct pathogenic evidence regarding the effects of diabetic control on the development of small fiber degeneration.

Neurotrophins are a gene family of structurally related proteins that is released by target tissues of responsive peripheral nerves, binds to specific receptors, and regulates gene expression through the actions of second-messenger systems. Each member of the family has its selectively tropical effects on peripheral nerves and plays a role in promoting neurite outgrowth, inducing morphological differentiation, stimulating expression and release of neurotransmitters and promoting nerve regeneration. It is hypothesized that abnormal availability of neurotrophins is involved in the pathogenesis of diabetic neuropathy. Studies have showed reduced seral level of neurotrophins in diabetic patients but it is not clear whether the impact of this finding on the diabetic neuropathy. There have no studies demonstrating if nay correlation between abnormal neurotrophins expression and the pathogenesis of small fiber neuropathy in diabetic patients.

Skin biopsy with quantification of intraepidermal nerve fibers (IENF) is a new pathological approach to study small fiber sensory neuropathy. By applying this technique with enzyme linked immunosorbent assay, we will clarify the following issues:

1. Changes in skin innervation of neurologically asymptomatic type 2 diabetic patient.
2. The influence of diabetic control on the development of small fiber neuropathy.
3. The effect of neurotrophins on the pathogenesis of small fiber neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients fulfilling the diagnosis of type 2 diabetes mellitus19 and receiving oral hyperglycemic agent or insulin treatment with regular follow-up at outpatient clinics, (2) neurologically asymptomatic, i.e. absence of subjective motor or sensory symptom, and absence of motor or sensory sign on neurological examinations, (3) absence of renal impairment or other systemic disease, (4) absence of bleeding tendency, obvious limb edema, poor cardiopulmonary function, acute symptoms of poor diabetic control or any other contraindication for skin biopsy.

Exclusion Criteria:

* Use of anti-coagulant; any causes with bleeding tendency; moderate to severe limb edema; history of poor wound healing; poor hygiene and poor care patients; uremia under dialysis.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Tsang Hsieh, PhD, Study Director — Department of Anatomy and Cell Biology, National Taiwan University College of Medicine; Department of Neurology, National Taiwan University Hospital.
Locations (1):
- Department of Anatomy and Cell Biology, National Taiwan University College of Medicine, Taipei, Taiwan